CLINICAL TRIAL: NCT05957198
Title: Assessment of the Oxygen Use and Future Outcomes Associated With Oxygen Use in Patient With Fibrotic ILD
Brief Title: Oxygen Therapy Use in Patients With Fibrotic Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0541
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with fibrotic interstitial lung disease (ILD): Patients aged ≥18 years with ≥2 fibrosing ILD diagnoses and continuous enrollment with medical and pharmacy coverage for 12 months prior to the fibrosing ILD diagnosis date as recorded in a commercial, Medicaid, or Medicare plan, using existing administrative claims and EHR data in Optum's Market Clarity Integrated Claims + Clinical database for the patient identification period (01-Oct-2016 through 30-Jun-2022).

SUMMARY:
The purpose of this study is to describe initiation and use of oxygen therapy among patients with fibrotic Interstitial Lung Disease (ILD) and to assess the impact of oxygen therapy on clinical outcomes among patients with fibrotic ILD.

ELIGIBILITY:
Inclusion criteria:

* ≥2 fibrosing Interstitial Lung Disease (ILD) diagnoses in any position on different dates of service, within 365 days of each other, and in the same continuous enrollment period during the patient identification period. The fibrosing ILD diagnosis date will be defined as the date of the first fibrosing ILD diagnosis. The two fibrosing ILD diagnosis codes can be one of the following combinations:
* 2 fibrosis codes
* 1 fibrosis code & 1 ILD code that requires fibrosis code
* ≥18 years of age as of the fibrosing ILD diagnosis date
* Continuous enrollment with medical and pharmacy coverage for 12 months prior to the fibrosing ILD diagnosis date (pre-ILD baseline period)

Exclusion criteria:

* Fibrosing ILD diagnosis in the 12-month pre-ILD baseline period
* Unknown gender, geographic region, or insurance type

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with fibrosing Interstitial Lung Disease (ILD) during the patient identification period.
Sampling Method: Probability Sample
Enrollment: 114921 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim Pharmaceuticals, Inc., Ridgefield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional study in patients with Fibrotic Interstitial Lung Disease (ILD) enrolled in a commercial, Medicaid, or Medicare plan, using existing administrative claims and Electronic Health Record (EHR) data in Optum's Market Clarity Integrated Claims + Clinical database for the period of 01 October 2015 through 30 June 2022 (study period). The patient identification period was (01-Oct-2016 through 30-Jun-2022).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial.
Period: Overall Study
Arm/Group | Patients With Fibrotic Interstitial Lung Disease (ILD)
Started | 114921
Completed | 114921
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients aged ≥18 years with newly diagnosed fibrosing ILD were identified from 01 October 2016 through 30 June 2022 (patient identification period) in existing data from a commercial, Medicaid, or Medicare plan, using existing administrative claims and electronic health record (EHR) data in Optum's Market Clarity Integrated Claims + Clinical database.
Arm/Group | Patients With Fibrotic Interstitial Lung Disease (ILD)
Number analyzed (Participants) | 114921
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60669
  Male | 54252
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5455
  Not Hispanic or Latino | 78150
  Unknown or Not Reported | 31316
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1824
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11492
  White | 77744
  More than one race | 0
  Unknown or Not Reported | 23861

OUTCOME MEASURES:

1. Primary Outcome: Time to Oxygen Therapy Initiation
Description: Time from the fibrosing Interstitial Lung Disease (ILD) diagnosis date to oxygen therapy initiation is reported.
  Descriptive statistics are rounded to one decimal place.
Time Frame: Up to 2099 days (from 01 October 2016 through 30 June 2022 (patient identification period)).
Population: Population AIM 1 include patients newly diagnosed with fibrosing ILD during the patient identification period and met all the eligibility criteria.
  Population AIM 1 in this endpoint restricted to patients without baseline oxygen therapy use.
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Idiopathic Pulmonary Fibrosis (IPF) Cohort: Patients aged ≥ 18 years with newly diagnosed fibrosing interstitial lung disease (ILD) during the patient identification period with ≥2 fibrosing ILD diagnoses, continuous enrollment with medical and pharmacy coverage for 12 months prior to the fibrosing ILD diagnosis date (pre-ILD baseline period) and ≥2 medical claims with diagnosis for idiopathic pulmonary fibrosis (IPF) in any position during the study period.
- Non Idiopathic Pulmonary Fibrosis (IPF) Cohort: Patients aged ≥ 18 years with newly diagnosed fibrosing interstitial lung disease (ILD) during the patient identification period with ≥2 fibrosing ILD diagnoses, continuous enrollment with medical and pharmacy coverage for 12 months prior to the fibrosing ILD diagnosis date (pre-ILD baseline period) and no claims with diagnosis for idiopathic pulmonary fibrosis (IPF) in any position during the study period.
Arm/Group | Idiopathic Pulmonary Fibrosis (IPF) Cohort | Non Idiopathic Pulmonary Fibrosis (IPF) Cohort
Number analyzed (Participants) | 4779 | 88799
Months | 27.5 [25.4 to 29.6] | NA [NA to NA] — Due to the insufficient number of events the median could not be calculated.

2. Primary Outcome: Sustained Oxygen Therapy Use Within the First 12 Months of Follow-up
Description: The number of participants with ≥ 11 claims for oxygen therapy within 12 months of initiating oxygen therapy is reported.
  Using claims, sustained oxygen therapy use was defined among patients with at least 12 months of follow-up after the index date (oxygen initiation date), as a binary variable for the presence of ≥11 claims for oxygen therapy in a 12-month period.
Time Frame: Up to month 12 of follow-up, in patient identification period from 01 October 2016 through 30 June 2022.
Population: Population AIM 1 include patients newly diagnosed with fibrosing ILD during the patient identification period and met all the eligibility criteria.
  Population AIM 1 in this endpoint restricted to patients with sustained oxygen therapy use within 12 months of initiating oxygen therapy patients and with ≥ 11 claims for oxygen therapy within 12 months of initiating oxygen therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Idiopathic Pulmonary Fibrosis (IPF) Cohort | Non Idiopathic Pulmonary Fibrosis (IPF) Cohort
Number analyzed (Participants) | 1339 | 10592
Participants | 967 | 4973

3. Primary Outcome: Time to Sustained Oxygen Therapy Use
Description: Time between the fibrosing ILD diagnosis date and the earliest date that defined the sustained oxygen therapy use is reported.
  Sustained oxygen therapy was defined as ≥ 11 claims for oxygen therapy within 12 months of initiating oxygen therapy.
Time Frame: Up to 2099 days (from 01 October 2016 through 30 June 2022 (patient identification period)).
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Idiopathic Pulmonary Fibrosis (IPF) Cohort | Non Idiopathic Pulmonary Fibrosis (IPF) Cohort
Number analyzed (Participants) | 967 | 4973
Days | 275 [184 to 305] | 266 [142 to 305]

4. Primary Outcome: Number of Participants With Disease Progression From Pre-index Forced Vital Capacity (FVC) Result to Index Date
Description: The Number of participants with disease progression is reported instead of time to disease progression in the Outcome Measure Data Table.
  Disease progression was defined as a 10% relative change between the forced vital capacity (FVC) pre-index value and the index date.
Time Frame: Up to 12 months prior to the index date (between 01 October 2016 through 30 June 2022 (patient identification period)).
Population: Among the 24,686 fibrosing Interstitial Lung Disease (ILD) patients who initiated oxygen therapy during the Aim 1 follow-up period, 24,680 were successfully matched at a 1:1 ratio with a fibrosing ILD patient who did not yet initiate oxygen therapy.
  Patients of the matched cohort are included for which pre-index and follow-up forced vital capacity (FVC) results were available.
Measure: Count of Participants; unit: Participants
Groups:
- Oxygen Use Cohort: Interstitial lung disease (ILD) patients with ≥1 medical claim for oxygen therapy after fibrosing ILD diagnosis.
- No Oxygen Use Cohort: Patients who were matched to a patient in the oxygen therapy cohort.
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Participants | 162 | 110

5. Primary Outcome: Number of Participants With Disease Progression From Index Date to Follow-up Forced Vital Capacity (FVC) Result
Description: The Number of participants with disease progression is reported instead of time to disease progression in the Outcome Measure Data Table.
  Disease progression was defined as a 10% relative change between the index date to follow-up FVC result.
Time Frame: Up to month 12 of follow-up, in patient identification period from 01 October 2016 through 30 June 2022.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Participants | 575 | 456

6. Primary Outcome: Time to All-cause Mortality
Description: Time to all-cause mortality is calculated as time between index date and mortality date.
  The oxygen therapy cohort index date was defined as the first date of a claim for oxygen therapy.
  The no oxygen therapy cohort index date was assigned as a date that was eligible to set an index date.
Time Frame: Up to 2099 days (from 01 October 2016 through 30 June 2022 (patient identification period)).
Population: Population AIM 2 include ILD patients with ≥1 medical claim for oxygen therapy after fibrosing ILD diagnosis of patients identified for AIM 1 and patients of AIM 1 who matched by propensity score matching (PSM) procedure.
  For each oxygen therapy cohort patient, a patient who had not yet initiated oxygen therapy and with the closest available propensity score was selected.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Months | 53.8 [50.8 to 56.5] | NA [NA to NA] — Due to the insufficient number of events the median could not be calculated.

7. Secondary Outcome: Percentage of Participants With Hypoxemia in the Pre-Interstitial Lung Disease (ILD) Baseline Period
Description: Percentage of participants with hypoxemia in the pre-ILD baseline period. The Percentage of participants is reported instead of time to hypoxemia in the Outcome Measure Data Table.
  The pre-ILD baseline period is defined as 12 months prior to the fibrosing ILD diagnosis date.
Time Frame: Up to 12 months prior to the fibrosing ILD diagnosis date (between 01 October 2016 through 30 June 2022 (patient identification period)).
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Percentage of Participants | 19.9 | 14.8

8. Secondary Outcome: Percentage of Participants With Hypoxemia in the Pre-index Baseline Period
Description: Percentage of participants with hypoxemia in the pre-index baseline period. The Percentage of participants is reported instead of time to hypoxemia in the Outcome Measure Data Table.
  The pre-index period was defined as the 12-month period prior to the index date. The index date is the first day of follow-up observation time for Aim 2.
Time Frame: Up to 12 months prior to the index date (between 01 October 2016 through 30 June 2022 (patient identification period)).
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Percentage of Participants | 57.2 | 21.0

9. Secondary Outcome: Percentage of Participants With Acute Exacerbations Within the First 12 Month of the Follow up Period
Description: Percentage of participants with acute exacerbations within the first 12 month of the follow up period. The Percentage of participants is reported instead of time to acute exacerbations in the Outcome Measure Data Table.
  The follow up period (variable period) started on the index date until the earliest of the following: disenrollment from the health plan, death, or the end of the study period.
Time Frame: Up to 12 months post index date (between 01 October 2016 through 30 June 2022 (patient identification period)).
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Percentage of Participants | 3.5 | 1.6

10. Secondary Outcome: Percentage of Participants With Acute Exacerbations in the Pre-index Baseline Period
Description: Percentage of participants with acute exacerbations in the pre-index baseline period. The Percentage of participants is reported instead of time to acute exacerbations in the Outcome Measure Data Table.
  The pre-index period was defined as the 12-month period prior to the index date. The index date is the first day of follow-up observation time for Aim 2.
Time Frame: Up to 12 months prior to the index date (between 01 October 2016 through 30 June 2022 (patient identification period)).
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Oxygen Use Cohort | No Oxygen Use Cohort
Number analyzed (Participants) | 24680 | 24680
Percentage of Participants | 2.8 | 1.3

ADVERSE EVENTS:
Time Frame: Not applicable for other Adverse Events (AEs) and serious AEs. All-Cause mortality was recorded between 01 October 2016 and 30 June 2022, up to 2099 days.
Description: This is a study with secondary use of data, safety reporting on an individual case level is not applicable. Other Adverse Events (AEs) and Serious AEs were not collected. "0" total Number of Participants at Risk means not collected.
  All-cause mortality is reported on AIM 1 population because AIM 2 does not include all subjects and deaths. AIM 1 is larger but it is not divided by oxygen use.
Arm/Group | Patients With Fibrotic Interstitial Lung Disease (ILD)
All-Cause Mortality (participants affected / at risk) | 21503/114921
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
* All ILD patients included in this study were enrolled in a health during the study period; thus, findings from this study may not be applicable to uninsured populations and patients with health plans not represented in the database.
* This study minimized bias by utilizing propensity score matching on baseline variables to examine outcomes of interest. Employing matching enabled a comparison of outcomes among patients who were similar on pre-ILD baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT05957198/Prot_SAP_000.pdf